CLINICAL TRIAL: NCT05379101
Title: Intracardiac Flow Assessment in Cardiac Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ian C. Chang, Principal Investigator, Mayo Clinic
Other Study IDs: 22-001098
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Amyloidosis Cardiac; Healthy Adults
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Echocardiography; Walk Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Transthyretin (ATTR) cardiac amyloidosis: Subjects diagnosed with ATTR cardiac amyloidosis will have CMR, TTE, and 6-minute walk
  Interventions: Diagnostic Test: Cardiac magnetic resonance image (CMR); Diagnostic Test: Transthoracic Echocardiogram (TTE); Diagnostic Test: Six-minute Walk Test
- Light chain amyloidosis (AL) with cardiac involvement: Subjects diagnosed with AL with cardiac involvement will have CMR, TTE, and 6-minute walk
  Interventions: Diagnostic Test: Cardiac magnetic resonance image (CMR); Diagnostic Test: Transthoracic Echocardiogram (TTE); Diagnostic Test: Six-minute Walk Test
- Light chain amyloidosis (AL) without cardiac involvement: Subjects diagnosed with AL without cardiac involvement will have CMR, TTE, and 6-minute walk
  Interventions: Diagnostic Test: Cardiac magnetic resonance image (CMR); Diagnostic Test: Transthoracic Echocardiogram (TTE); Diagnostic Test: Six-minute Walk Test
- Healthy Control: Subjects without history of cardiovascular diseases will have CMR, TTE, and 6-minute walk
  Interventions: Diagnostic Test: Cardiac magnetic resonance image (CMR); Diagnostic Test: Transthoracic Echocardiogram (TTE); Diagnostic Test: Six-minute Walk Test

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance image (CMR) — A magnetic resonance imaging study for assessment of cardiac structure and intracardiac flow
Diagnostic Test: Transthoracic Echocardiogram (TTE) — An imaging test that uses soundwaves that cannot be heard (ultrasound) to take pictures of the heart and vessels.
Diagnostic Test: Six-minute Walk Test — A self-paced, test of exercise capacity performed unencouraged intensity that measures the distance that patients can walk on a flat, hard surface in a period of 6 minutes

SUMMARY:
The primary objective of this study is to define the intracardiac flow imaging biomarkers in cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is clinically stable without cardio-vascular-related hospitalizations within 6 weeks prior to enrollment as assessed by the investigators.
* Subject is able to provide written informed consent and is willing and able to complete study procedures.
* Currently in sinus rhythm by clinical assessment or documented electrocardiographic studies.
* Subject and disease characteristics noted by medical record review:

  * Healthy control volunteers must also meet the following criteria: Karnofsky performance scale > 80%; ECOG status 0 or 1.
  * ATTR cardiac amyloidosis based on meeting all the following criteria: Diagnosis of amyloidosis within five years prior to study screening; Documentation of absence of AL, heavy chain disease, multiple myeloma or malignant lymphoproliferative disorders; Transthyretin amyloid deposits in cardiac tissue OR technetium (99mTc) pyrophosphate scintigraphy with grade 2 or 3 cardiac uptake OR Transthyretin amyloid deposits in non-cardiac tissue with echocardiographic evidence of cardiac involvement or an end-diastolic mean wall thickness >12mm OR Transthyretin amyloid deposits in non-cardiac tissue with CMR diagnostic of amyloidosis
  * AL with cardiac involvement based on meeting all the following criteria: Diagnosis of amyloidosis within five years prior to study screening; Histopathologic diagnosis of amyloidosis with AL protein identification; Documented clinical signs or symptoms consistent with heart failure; Cardiac involvement as defined by: Amyloid deposits in cardiac deposits OR Echocardiography with an end-diastolic mean wall thickness > 12 mm in the absence of other causes OR Elevated NT-proBNP (>332 ng/L) in the absence of renal failure or atrial fibrillation OR CMR diagnostic of amyloidosis;
  * AL without cardiac involvement based on meeting all the following criteria: Diagnosis of amyloidosis within five years prior to study screening; Histopathologic diagnosis of amyloidosis with AL protein identification; No documented clinical signs and symptoms consistent with heart failure from AL; Absence of cardiac involvement as defined by: Echocardiography with an end-diastolic mean wall thickness < 13 mm if the subject does not have other causes for increased wall thickness AND NT-proBNP <333 ng/L if the subject does not have renal failure or atrial fibrillation AND No CMR diagnostic of amyloidosis if CMR is available prior to screening.

Exclusion Criteria:

* Unable to consent or unable to complete all study procedures.
* Unable to ambulate for 6 minutes (confirmed at study coordinator visit).
* Unable to maintain in supine position for 30 minutes.
* Unable to maintain breath-holding for 10 seconds (confirmed at study coordinator visit).
* Contraindications for safe CMR scanning (e.g., uncontrolled claustrophobia, cochlear implant, implanted neural stimulator).
* Presence of implantable cardiac pacemaker or defibrillator.
* History of complex congenital heart disease, intracardiac shunt (except for patent foramen ovale), prosthetic valves, prosthesis in the main pulmonary artery or ascending thoracic aorta.
* Significant artifact from prior MRI studies.
* Pregnant or breast-feeding women.
* Weight equal to or greater than 155 kg.
* Maximum body side-to-side or anterior-posterior diameter equal to or greater than 70 cm.
* Documented non-sinus rhythm within 1 week prior to screening.
* For healthy controls, the following exclusion criteria apply, confirmed per chart review and/or patient report:

  * History of cardiomyopathy or structural heart disease;
  * History of valvular disease of greater than mild severity;
  * History of coronary artery disease or coronary heart disease;
  * History of cardiac or thoracic surgery.
  * History of symptomatic, persistent atrial tachyarrhythmia, ventricular tachyarrhythmia, or bradyarrhythmia;
  * Left ventricular hypertrophy or abnormally increased myocardial thickness by prior echocardiography, cardiac computed tomography, or CMR;
  * Acute kidney injury, OR chronic renal disease with glomerular filtration rate < 45 mL/min/1.73m^2 as per medical record review.
  * Uncontrolled hypertension of systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg as per medical record review;
  * Taking three or more anti-hypertensive medications;
  * Type 1 diabetes, OR uncontrolled type 2 diabetes mellitus of hemoglobin A1c greater than 8, as per medical record review;
  * Taking three or more diabetic medications;
  * History of confirmed stroke or transient ischemic attack, as per medical record review;
  * Current cigarette smoker;
  * History of plasma cell dyscrasia or chronic malignant hematologic diagnosis;
  * BMI > 35 kg/m^2.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with amyloidosis without and with cardiac involvement, and normal healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Define the intracardiac flow imaging biomarkers in cardiac amyloidosis (CA) | Baseline
  Measured by cardiac magnetic resonance imaging (CMR)

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Chang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No